CLINICAL TRIAL: NCT03837236
Title: Inactivity Behavior and Exercise Bariers in Patients With Behçet Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Behçet Disease
Keywords: Behçet disease; Physical activity level; Exercise barriers
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Evaluation parameters will be performed to the patients. Physical activity level, exercise barriers, disease activity, fatigue, depression, pain, sleep disorders, aerobic capacity and quality of life will be assessed using International Physical Activity Questionnaire-Short Form (IPAQ),Exercise Benefits/Barriers Scale, Behçet Disease Current Activity Form (BDCAF), Fatigue Severity Scale (FSS), Beck Depression Inventory (BDI), McGill Pain Questionnaire- Short Form (MPQ-SF), Pittsburgh Sleep Quality Index, 6 minute walk test and Behçet's Disease Quality of Life Questionnaire, respectively.
  Interventions: Other: Study group

INTERVENTIONS:
Other: Study group — Evaluation parameters will be performed to the patients. Physical activity level, exercise barriers, disease activity, fatigue, depression, pain, sleep disorders, aerobic capacity and quality of life will be assessed using International Physical Activity Questionnaire-Short Form (IPAQ),Exercise Benefits/Barriers Scale, Behçet Disease Current Activity Form (BDCAF), Fatigue Severity Scale (FSS), Beck Depression Inventory (BDI), McGill Pain Questionnaire- Short Form (MPQ-SF), Pittsburgh Sleep Quality Index, 6 minute walk test and Behçet's Disease Quality of Life Questionnaire, respectively.

SUMMARY:
Behçet's Disease (BD) is a chronic, inflammatory, rheumatic disease that is characterized by mucocutaneous lesions. Promoting physical activity level is one of the major goals in the management of patients with rheumatic diseases, it is important to determine the factors affecting physical activity level and exercise barriers. The aim of this study is to investigate physical activity level and exercise barriers in patients with BD. Physical activity level, exercise barriers, disease activity, fatigue, depression, pain, sleep disorders, aerobic capacity and quality of life will be assessed using International Physical Activity Questionnaire-Short Form (IPAQ),Exercise Benefits/Barriers Scale, Behçet Disease Current Activity Form (BDCAF), Fatigue Severity Scale (FSS), Beck Depression Inventory (BDI), McGill Pain Questionnaire- Short Form (MPQ-SF), Pittsburgh Sleep Quality Index, 6 minute walk test and Behçet's Disease Quality of Life Questionnaire, respectively.

DETAILED DESCRIPTION:
Behçet's Disease (BD) is a chronic, inflammatory, rheumatic disease that is characterized by mucocutaneous lesions and can be seen major organ involvement such as eyes, musculoskeletal system, gastrointestinal system and central nervous system. Gender and clinical findings effect the prognosis of the disease. Physical activity is all body movements requiring energy expenditure over basal metabolism and contraction of skeletal muscle. Promoting physical activity level is one of the major goals in the management of patients with rheumatic diseases because of negative impact of sedentary lifestyle which depends on rheumatic involvement.Impaired quality of life, aerobic capacity, respiratory function and life satisfaction, sleep disorders, depression, anxiety and fatigue are seen commonly in BD patients like the other rheumatic diseases. Because of these symptoms, it is possible and expected that BD patients have low physical activity level. Considering that regular physical activity effects survival for patients and healthy people, it is important to determine the factors affecting physical activity level and exercise barriers. The aim of this study is to investigate physical activity level and exercise barriers in patients with BD. Physical activity level, exercise barriers, disease activity, fatigue, depression, pain, sleep disorders, aerobic capacity and quality of life will be assessed using International Physical Activity Questionnaire-Short Form (IPAQ),Exercise Benefits/Barriers Scale, Behçet Disease Current Activity Form (BDCAF), Fatigue Severity Scale (FSS), Beck Depression Inventory (BDI), McGill Pain Questionnaire- Short Form (MPQ-SF), Pittsburgh Sleep Quality Index, 6 minute walk test and Behçet's Disease Quality of Life Questionnaire, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Being followed at the Gazi University Faculty of Medicine, Department of Rheumatology with Behçet Disease met the diagnostic criteria proposed at the International Study Group of Behçet Disease.
* The age of 18- 65 years

Exclusion Criteria:

* Illiterate,
* Pregnant
* Diagnosed with malignancy
* Accompaning any other rheumatic diseases except from Fibromyalgia
* Having changes of medical treatment in the last 3 months
* having dysfunction that limited physical activity such as severe neurological impairment, immobility or cooperation deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-05-08 (Estimated); Study Completion 2019-11-08 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ)- Short Form | 1 minute
  This questionnaire obtains information about how much time is spent while walking and in moderate and vigorous activities and sitting duration in the last 7 days. The questionnaire records the activity of four intensity levels: 1) vigorous-intensity activity, 2) moderate-intensity activity, 3) walking, and 4) sitting. Durations are multiplied by known METs per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. A sitting question is not included in physical activity score. The questionnaire is scored as: those who score high on the IPAQ engage in vigorous intensity activity of at least 1500 MET minutes a week, those who score modarete on the IPAQ of at least 600 MET minutes a week, those who score a low level of physical activity on the IPAQ means that not meeting any of the criteria for either moderate or high levels of physical activity.
the Exercise Benefits/Barriers Scale | 2 minutes
  It consists of 43 items including benefits of exercise (e.g. I enjoy exercise) and barriers (e.g. Exercising takes too much of my time). Benefits subscale scores range between 29 and 116 while barriers subscale scores range between 14 and 56. The higher the score on the Barriers scale, the greater the perception of barriers to exercise.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 2 minutes
  This scale consists of nine questions; each question is scored from 1 to 7, in which a high FSS score indicates severe fatigue.
Beck Depression Inventory | 1 minute
  Beck Depression Inventory consists of 21 items related to depressive symptoms such as pessimism, sense of failure, guilt, dissatisfaction, sleep, appetite and fatigue. Each item is scored between 0 and 3. Higher score means increased severity of depression. According to this scale 1-10 points are defined as normal, scores between 11-16 indicate mild mental distress, 17-20 indicate the patient is at the border points for clinical depression, 21-30 indicate moderate depression, severe depression scores are between 31-40 and 40 points above are interpreted as a very serious depression.
Short Form McGill Pain Questionnaire | 2 minutes
  This questionnaire consists of 11 sensory and 4 affective descriptive words. These 15 words are scored range between 0 and 4. So three type of pain scores (sensory, affective, total = sensory + affective) are obtained. In McGill Pain Questionnaire, the current level of pain is measured by Visual Analog Scale (VAS) and Likert scale consisting of 6 points (0 = no pain, 1 = mild, 2 = irritating, 3 = bothersome, 4 = terrible, 5 = unbearable).
Behçet's Disease Quality of Life Questionnaire | 5 minutes
  It consists of 15 items about difficulties in social, psychological and daily living effects for patients with BD. All questions have the same five answers including; always (4 points), usually (3 points), sometimes (2 points), rarely (1 point), never (0 point). Total score is calculated by collecting all points, which ranges between 0 and 60 points. The higher score indicated the high quality of life level.
Pittsburgh Sleep Quality Index | 2 minutes
  It is a self-assessment questionnaire which evaluates sleep quality and disturbances over a 1 month time interval. It consists of 19 self-rated items and five questions rated by the bedpartner or roommate which is not included to the total score. . These 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component scores are then summed yo yield a global Pittsburgh Sleep Quality Index score, which has a range of 0-2 and the higher score indicates worse sleep quality.
6 minute walk test | 6 minutes
  6MWT is a distance required to fast-paced walk on flat floor in length 30 meters. The aim of the 6MWT is to walk as long as the patient can walk in 6 minutes. Dyspnoea and fatigue level are recorded at the end of the test.
Behçet Disease Current Activity Form (BDCAF) | 5 minutes
  It has 12 components; headache, oral ulcer, genital ulcer, arthralgia, erythema, skin pustule, arthritis, nausea/vomiting/abdominal pain, diarrhea or frank blood per rectum, eye symptoms, nervous and vascular system symptoms. Each component is scored as absent (0 point) or present (1 point) and final BDCAF score is sum of all components with a maximum of 12.

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Study Director — Gazi University Faculty of Health Sciences
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moses Alder N, Fisher M, Yazici Y. Behcet's syndrome patients have high levels of functional disability, fatigue and pain as measured by a Multi-dimensional Health Assessment Questionnaire (MDHAQ). Clin Exp Rheumatol. 2008 Jul-Aug;26(4 Suppl 50):S110-3. PMID 19026127
- [Result] Hatemi G, Merkel PA, Hamuryudan V, Boers M, Direskeneli H, Aydin SZ, Yazici H. Outcome measures used in clinical trials for Behcet syndrome: a systematic review. J Rheumatol. 2014 Mar;41(3):599-612. doi: 10.3899/jrheum.131249. Epub 2014 Feb 1. PMID 24488418